CLINICAL TRIAL: NCT02578082
Title: The Effect of Severe Renal Impairment on the Pharmacokinetics Following Single-Dose Inhaled Administration of TD 4208
Brief Title: Pharmacokinetics of TD-4208 in Patients With Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0135
Record Dates: First submitted 2015-10-08; First posted 2015-10-16 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Renal Impairment
Keywords: Renal Impairment; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — revefenacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal Impairment (Experimental): Eight subjects with Severe Renal Impairment (eGFR <30 mL/min/1.73m2). Intervention is TD-4208, 175mcg, inhaled, single dose.
  Interventions: Drug: TD-4208
- Normal Renal Function (Experimental): Eight healthy participants matched to participants with severe renal impairment.
  Intervention is TD-4208, 175mcg, inhaled, single dose.
  Interventions: Drug: TD-4208

INTERVENTIONS:
Drug: TD-4208 — A single inhaled dose of TD 4208 (175 mcg)
  Other Names: revefenacin

SUMMARY:
This multiple-center, nonrandomized, open label, parallel group, single dose study will be conducted in male and female subjects with normal renal function or severe (eGFR <30 mL/min/1.73 m2) renal impairment to evaluate the effect of renal impairment on the pharmacokinetics (PK) of TD 4208.

ELIGIBILITY:
Inclusion Criteria:

For renal impairment group:

* Subject has severe renal impairment (eGFR <30 mL/min/1.73 m2)

For normal renal function group:

* Subject is in good health

Exclusion Criteria:

* Women who are pregnant, lactating, breastfeeding, or planning to become pregnant during the study.
* Subject has received an investigational drug (or medical device) within 30 days
* Subject who, for any reason, is deemed by the investigator to be inappropriate for this study; or has any condition that would confound or interfere with the evaluation of the safety, tolerability, or PK of the investigational drug; or is unable to comply with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Predose; 5min, 15min, 30 min; 1hr, 2hr, 3hr, 4hr, 6hr, 8hr, 12hr, 24hr, 36hr, 48hr, 72hr, 96hr post dose
  TD-4208 Cmax derived from plasma concentration-time curves

SECONDARY OUTCOMES:
Adverse Events (AE) | From the time of study drug administration through the end of the study (Day 5 or early termination)
  An AE is any unfavorable and unintended change in the body temporally associated with study drug administration, whether or not considered related to the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Orlando Clinical Research Center (OCRC), Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borin MT, Lo A, Barnes CN, Pendyala S, Bourdet DL. Pharmacokinetics and safety of revefenacin in subjects with impaired renal or hepatic function. Int J Chron Obstruct Pulmon Dis. 2019 Oct 8;14:2305-2318. doi: 10.2147/COPD.S203709. eCollection 2019. PMID 31632000